CLINICAL TRIAL: NCT05879159
Title: Accelerated Recovery After MIS Hepatectomy (ARAMIS Hep) to Support Early Discharge for Patients Undergoing Minimally Invasive Liver Resection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Intuitive Surgical Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-0917; NCI-2023-04169 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Liver
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accelerated Recovery Protocol (Experimental): Accelerated Recovery after Minimally Invasive Hepatic Surgery (ARAMIS-Hep)
  Participants randomized to this arm will undergo a recovery pathway that potentially allows for discharge on the day of surgery (post-operative day 0).
  * You will receive a clear liquid diet, be encouraged to ambulate independently, and opioid use will be minimized in the recovery unit.
  * You will be assessed in the post-operative recovery unit. If you meet discharge criteria, you will be discharged the afternoon/evening of surgery. If you do not, you will be admitted for overnight observation.
  * You will have a telehealth video visit on post-operative days 1 and 2
  * You will have in-person clinic visit within 14 days of discharge.
  You will fill out about 14 questionnaires over a 30-day period to assess how you are feeling regarding your recovery
  Interventions: Behavioral: Questionnaires
- Comparison/Control Arm (Experimental): Standard Post-operative recovery pathway after minimally invasive hepatic surgery.
  Participants randomized to this arm will undergo our institution's standard recovery pathway for minimally invasive liver surgery.
  * You will be transferred to the Transitional PACU for overnight observation.
  * Your diet will be advanced to gastrointestinal "first food" diet on Post-operative Day 1, with opioid weaning and frequent ambulation.
  * You will be discharged once criteria are met.
  * You will have an in-person clinic visit within 14 days of discharge.
  You will fill out about 14 questionnaires over a 30-day period to assess how you are feeling regarding your recovery.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Survey

SUMMARY:
To learn if an accelerated recovery program can shorten the length of hospital stay in patients having minimally invasive liver surgery.

DETAILED DESCRIPTION:
Primary Objectives:

Our study will investigate the feasibility of an accelerated recovery program to minimize length of stay (LOS) and facilitate outpatient surgery for patients undergoing minimally invasive, lower complexity (Kawaguchi-Gayet grade I) liver resection. This program (ARAMIS Hep) will combine minimally invasive surgical (MIS) approaches (robotic OR laparoscopic), enhanced recovery after surgery (ERAS) protocols, and Telehealth to liberalize discharge criteria in a safe manner.

Secondary Objectives:

In addition to demonstrating a reduction in LOS, our study will also provide preliminary data to aid in the broader implementation of this approach. Specifically, we will gain insight into the patient experience, measure patient-reported outcomes on recovery trajectories, and understand barriers to integrating a novel pathway into existing institutional frameworks.

ELIGIBILITY:
Inclusion Criteria:

* Tumor amenable to MIS Kawaguchi-Gayet grade I hepatectomy (see figure 1 below)
* No evidence of cirrhosis (based on imaging, evidence of portal hypertension, clinical features, or laboratory results)
* No significant cardiopulmonary disease that would prevent patients from undergoing MIS resection
* Ability to stay within 50 miles of medical center for immediate postop period
* Age of 18 years or above - because no adverse event data are currently available on enhanced recovery and early discharge after hepatic resection for patients <18 years of age, children are excluded from this study
* Ability to understand and the willingness to sign a written informed consent document
* Non-English-speaking patients are eligible for participation

Exclusion Criteria:

Patients who will be excluded include those with:

* Tumors NOT amenable to MIS Kawaguchi-Gayet grade I hepatectomy
* Tumors not amenable to MIS or Robotic-assisted surgical resection
* Evidence of Cirrhosis on imaging, clinically, or lab testing
* Inability to stay within 50 miles of the Cancer Center in the immediate post-operative period
* Age below 18 years
* Inability to consent for trial/protocol
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Hop Tran Cao, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org